CLINICAL TRIAL: NCT03462069
Title: A Randomized, Double-blind, Parallel-group, 2-treatment Multiple Dose Study to Assess the Intestinal, Metabolic and Cardiovascular Effects of an 8 Weeks Treatment With Sotagliflozin QD as Compared With Empagliflozin Once a Day (QD) in Type 2 Diabetes Mellitus (T2DM) Patients With Mild to Moderate Hypertension
Brief Title: Comparison of Pharmacodynamic Effects of Sotagliflozin and Empagliflozin in T2DM Patients With Mild to Moderate Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PDY15010; 2017-002309-36 (EudraCT Number); U1111-1186-2962 (Other: UTN)
Record Dates: First submitted 2018-03-06; First posted 2018-03-12 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — (2S,3R,4R,5S,6R)-2-(4-chloro-3-(4-ethoxybenzyl)phenyl)-6-(methylthio)tetrahydro-2H-pyran-3,4,5-triol; empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment A (Test) (Experimental): Sotagliflozin 2 tablets administered once daily with 1 empagliflozin placebo capsule prior to the first meal of the day
  Interventions: Drug: Sotagliflozin (SAR439954); Drug: Placebo
- Treatment B (Reference) (Active Comparator): Empagliflozin 1 capsule administered once daily with 2 sotagliflozin placebo tablets prior to the first meal of the day
  Interventions: Drug: Placebo; Drug: Empagliflozin

INTERVENTIONS:
Drug: Sotagliflozin (SAR439954) — Pharmaceutical form: tablet
  Route of administration: oral
  Arms: Treatment A (Test)
Drug: Placebo — Pharmaceutical form: tablet
  Route of administration: oral
  Arms: Treatment B (Reference)
Drug: Empagliflozin — Pharmaceutical form: capsule
  Route of administration: oral
  Other Names: Jardiance®
  Arms: Treatment B (Reference)
Drug: Placebo — Pharmaceutical form: capsule
  Route of administration: oral
  Arms: Treatment A (Test)

SUMMARY:
Primary Objective:

To compare the metabolic and gastrointestinal pharmacodynamic (PD) effects of an 8 weeks treatment with sotagliflozin once daily (QD) to an 8 weeks treatment to empagliflozin QD in mild or moderate hypertensive T2DM patients on a stable treatment regimen with metformin and an angiotensin converting enzyme (ACE) inhibitor or Angiotensin Receptor Blocker (ARB) under standardized diet conditions.

Secondary Objectives:

* To compare the renal and cardiovascular PD effects of an 8 weeks treatment with sotagliflozin QD to an 8 weeks treatment to empagliflozin QD in mild or moderate hypertensive T2DM patients on a stable treatment regimen with metformin and an ACE inhibitor or ARB.
* To evaluate the safety and tolerability of an 8 weeks QD treatment with sotagliflozin or empagliflozin in mild to moderate hypertensive T2DM patients on a stable treatment with metformin and an ACE inhibitor or ARB.
* To evaluate the pharmacokinetic (PK) profile of sotagliflozin in steady state conditions.

DETAILED DESCRIPTION:
The total study duration per patient is 70-105 days (for patients without drug washout/switch period), and up to 175 days (for patients with drug washout/switch period), including 2-30 days of screening, 5 days of run-in period, 56 days of treatment period, and a 7-14 days of follow-up period.

ELIGIBILITY:
Inclusion criteria :

* Male or female patients with Type 2 Diabetes Mellitus (T2DM) (diagnosed at least 1 year before screening visit), between 18 and 74 years of age, inclusive, with:

  * Hypertension grades 1 or 2 as defined by the European Society of Hypertension (ESH)/European Society of Cardiology (ESC) at screening; systolic blood pressure (SBP) has to be in the range of 140-179 mmHg (after 10 minutes resting in supine position, measurement in triplicate with each measurement to be within this range at screening). If the blood pressure (BP) range is not met at screening, one repeat measurement at another occasion is allowed prior to inclusion into the study.
  * Glycated Haemoglobin A1c (HbA1c) at screening between 6.5% and 11%.
* On a stable treatment with metformin, i.e., no change in dose regimen or in dose levels in the last 3 months prior to screening and throughout the study.
* On a stable treatment with an angiotensin converting enzyme (ACE) inhibitor or an angiotensin receptor blocker, i.e., no change in dose regimen or in dose levels in the last 4 weeks prior to screening and until randomization.
* On a stable treatment with an ACE inhibitor or an angiotensin receptor blocker after switching from beta-blockers and/or thiazides for eligible patients after screening, i.e., no change in dose regimen and in dose levels in the last 4 weeks prior to run-in phase and until randomization
* Body weight between 50.0 kg and 130 kg, inclusive, if male, and between 40.0 kg and 110 kg, inclusive, if female, body mass index between 18.0 and 38.0 kg/m2, inclusive.
* Kidney function: Estimated glomerular filtration rate at screening must be 60 mL/min/1.73m2 or higher.

Exclusion criteria:

* Patients with severe anemia, severe cardiovascular, gastrointestinal, respiratory, neurological, osteomuscular, psychiatric, or active malignant tumor or other major systemic disease or patients with infectious disease, signs of acute illness, or short life expectancy making implementation of the protocol or interpretation of the study results difficult (as evaluated by detailed medical history and complete physical and laboratory examination).
* Heart failure New York Heart Association (NYHA) Classification III/IV.
* Any clinically significant abnormality in echocardiography performed at screening as judged by the investigator based on age, gender and medical history of the individual patient.
* History of myocardial infarction within the last 12 months prior to screening.
* Likelihood of requiring treatment during the study period with drugs not permitted by the study protocol (e.g., long-term systemic glucocorticoids) and refusing or unable to take alternative treatment.
* Type 1 diabetes mellitus.
* Secondary hypertension of any etiology (eg, renovascular disease, pheochromocytoma, Cushing's syndrome).
* Clinically significant pulmonary hypertension, in particular World Health Organisation (WHO) Classes IV (Pulmonary hypertension due to chronic thrombotic and/or embolic disease [CTEPH]) and V (miscellaneous).
* Diabetic retinopathy.
* History of diabetic ketoacidosis or non-ketotic hyperosmolar coma within 12 weeks prior to the Screening Visit.
* History of severe hypoglycemia resulting in hospitalization or unconsciousness/seizures within 6 months prior to the Screening visit.
* History of prior gastric or intestinal surgical procedure including gastric banding within 3 years before the Screening Visit. Any gastrointestinal surgery with removal of part of the bowels or the stomach
* History of unexplained pancreatitis, chronic pancreatitis, stomach/gastric surgery, inflammatory bowel disease.
* Known hypersensitivity to sotagliflozin, empagliflozin or any excipient of the drug products.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-04-18 (Actual)

PRIMARY OUTCOMES:
Assessment of pharmacodynamic (PD) parameters in feces | Baseline and on Day 55 and 56 (over 48 hours)
  Change from baseline in fecal sodium excretion
Assessment of pharmacodynamic (PD) parameters in feces | Baseline and on Day 55 and 56 (over 48 hours)
  Change from baseline in fecal short-chain fatty acids (SCFA)
Assessment of pharmacodynamic (PD) parameters in feces | Baseline and on Day 55 and 56 (over 48 hours)
  Change from baseline in fecal pH
Assessment of PD parameters in urine | Baseline and on Day 56 (over 24 hours)
  Change from baseline in 24-hour urinary glucose excretion
Assessment of PD parameters in urine | Baseline and on Day 56 (over 24 hours)
  Change from baseline in 24-hour sodium excretion
Assessment of PD parameters in blood | Baseline and on Day 56
  14 hour plasma glucose profile after standardized meals
Assessment of PD parameters in blood | Baseline and on Day 56
  14 hour plasma glucagon-like peptide 1 (GLP-1) profile after standardized meals

SECONDARY OUTCOMES:
Fasting metabolic laboratory panel | Baseline and on Day 56
  Change from baseline in fasting plasma glucose
Ambulatory Blood Pressure Measurement (ABPM) | Baseline and on days 54 until Day 56
  Change from baseline in average 24h systolic arterial pressure
Cardiovascular parameters | Baseline and on Day 56
  Change from baseline in plasma aldosterone
Pulse wave velocity | Baseline and on Day 55
  Change from baseline in carotid-femoral pulse wave velocity
Continuous Glucose Monitoring (CGM) | Baseline, last 3 days of treatment
  Change from baseline in average diurnal glucose
Echocardiography | Baseline and on Day 54
  Change from baseline in left ventricular ejection fraction (LVEF)
Echocardiography | Baseline and on Day 54
  Change from baseline in left ventricular end-diastolic diameter
Plasma Volume Measurement | Baseline and on Day 54
  Change from baseline in plasma volume
Adverse events | Over 15 weeks
  Number of patients with reported adverse events
Assessment of pharmacokinetic (PK) parameters: Cmax | 24 hours after last investigational medicinal product (IMP) administration
  Sotagliflozin: maximum plasma concentration observed (Cmax)
Assessment of pharmacokinetic (PK) parameters: Ctrough | 24 hours after last IMP administration
  Sotagliflozin: plasma concentration observed before administration during repeated dosing (Ctrough)
Assessment of pharmacokinetic (PK) parameters: AUCtau | 24 hours after last IMP administration
  Sotagliflozin: Area under the plasma concentration versus time curve calculated using the trapezoidal method over the dosing interval (AUCtau)
Assessment of pharmacokinetic (PK) parameters: tmax | 24 hours after last IMP administration
  Sotagliflozin: First time to reach Cmax (tmax)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 2760001, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Posch MG, Walther N, Ferrannini E, Powell DR, Banks P, Wason S, Dahmen R. Metabolic, Intestinal, and Cardiovascular Effects of Sotagliflozin Compared With Empagliflozin in Patients With Type 2 Diabetes: A Randomized, Double-Blind Study. Diabetes Care. 2022 Sep 1;45(9):2118-2126. doi: 10.2337/dc21-2166. PMID 35817022